CLINICAL TRIAL: NCT06875206
Title: Visual Restoration Using Focused Ultrasound Stimulation and Immersive Virtual Reality After Stroke
Acronym: LIFU-IVR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00115941
Record Dates: First submitted 2025-02-11; First posted 2025-03-13 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Visual Field Defect; Visual Field Defect Following Cerebrovascular Accident; Hemianopia; Quadrantanopia; Occipital Lobe Infarct; Visual Fields Hemianopsia
Keywords: virtual reality; stroke; visual deficit; chronic stroke; ultrasound stimulation; neuromodulation; stroke recovery; visual field defect; funcational imaging
MeSH Terms: conditions — Stroke; Hemianopsia; Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LIFUS with IVR (Experimental): Participants are randomized to the active group will undergo active Low intensity-focused ultrasound stimulation (LIFUS) combined with Immersive Virtual Reality (IVR) therapy.
  Interventions: Device: Low-intensity focused ultrasound; Device: Immersive virtual reality
- Inactive LIFUS with IVR (Sham Comparator): The participants in the Sham group will undergo inactive low-intensity focused ultrasound stimulation combined with Immersive virtual reality therapy
  Interventions: Device: Immersive virtual reality; Device: Inactive Low-intensity focused ultrasound

INTERVENTIONS:
Device: Low-intensity focused ultrasound — Low-intensity focused Ultrasound (LIFU) is a noninvasive brain stimulation technique that uses low-intensity ultrasound to stimulate specific parts of the brain.
  Other Names: LIFU
  Arms: LIFUS with IVR
Device: Immersive virtual reality — IVR is a noninvasive, computer-based audiovisual therapy designed to enhance visual function. Using a VR headset, the system delivers targeted visual stimulation through an interactive game that the participant engages with during each session.
  Other Names: IVR
Device: Inactive Low-intensity focused ultrasound — High acoustic impedance disk placed between LIFU and scalp that mimics the audible sensation of a slight buzzing but attenuates more than 95% of the energy into the brain.
  Arms: Inactive LIFUS with IVR

SUMMARY:
This research will explore if brain stimulation combined with virtual reality therapy improves visual impairment. The stimulation technique is called low-intensity focused ultrasound stimulation (LIFUS). The treatment uses ultrasound to stimulate vision specific parts of the brain. Before this therapy, the participants will get structural brain imaging. Functional brain imaging will be performed before and after the study's completion to measure brain activity response to therapy.

The purpose of this research study is to evaluate patients who have had a stroke between 6 and 24 months ago with a visual field impairment. The duration of active participation in the study is 1.5 months.

DETAILED DESCRIPTION:
Randomization visit and 1st Intervention visit:

The randomization visit and 1st intervention vision will be on the same day. Participants will be "randomized" into one of the study groups described below.

* Group 1 (Sham Group): Inactive LIFU + VR
* Group 2 (Active Group): LIFU + VR Neither the subject nor the researcher conducting this study will know which group participants are in.

Sham LIFU: The setup is similar for the active stimulation group, except that a high acoustic impedance disk will be placed between the LIFU probe and the scalp that mimics the audible sensation of a slight buzzing but attenuates more than 95% of the energy into the brain. The audible sound is nearly identical for both the sham and active stimulation.

Intervention visits (9 sessions over 21 days, about 2.5 hours per visit):

At these visits, participants will undergo the investigational study interventions.

There will be 30 minutes of a VR session and 20 minutes of active LIFU or inactive LIFU treatments.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old of any gender and race
* Clinical ischemic stroke or hemorrhagic (confirmed by CT or MRI) that occurred >= 6-24 months ago
* Partial or complete homonymous hemianopsia on clinical exam

Exclusion Criteria:

* Documented history of severe dementia with or without medication before stroke that affect subject's ability to participate in and be compliant to study protocol
* Significant upper motor deficits and the subject cannot do IVR sessions at the baseline
* History of seizures
* Inability to get a new MRI
* Presence of any ultrasonic stimulation risk factors: an electrically, magnetically, or mechanically activated metal or nonmetal implant including cardiac pacemaker, intracerebral vascular clips, or any other electrically sensitive support system; non-fixed metal in any part of the body; pregnancy (the effect of ultrasonic stimulation on the fetus is unknown); preexisting scalp lesion or wound or bone defect or hemicraniectomy.
* Patients will be excluded if they have a previous diagnosis of hemianopsia, a new diagnosis of central retinal ischemic injury, or visual blindness or a history of any other ocular disease.
* Concerns about the inability to complete study visits/procedures by the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Visual Field Change | From enrollment to the 30 days after the end of treatment.
  Change of the blind area in the visual fields as measured by visual perimetry implemented in a virtual reality (VR) headset

SECONDARY OUTCOMES:
Quality of Life Change | From enrollment to the 30 days after the end of treatment.
  Change as assessed by the National Eye Institute 25 Item Visual Function Questionnaire (NEI-VFQ 25). The NEI-VFQ is a vision based questionnaire which evaluates quality of life with respect to vision in everyday life. The NEI-VFQ has multiple sub-scales for different areas of life, such as Near-Vision, General Health, or Ocular Pain. Each scale is scored from 0 to 100 with 100 representing the best possible score (perfect health or ability)
Hemodynamic response change | From enrollment to the 30 days after the end of treatment.
  Change in oxygenated hemoglobin concentration or blood-oxygen-level-dependent (BOLD) signal response from baseline and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No